CLINICAL TRIAL: NCT03227653
Title: Neuropsychiatric Adverse Effects of Efavirenz in Children Living With HIV in Kilimanjaro, Tanzania
Brief Title: Neuropsychiatric Side Effects of Efavirenz in Children Living With HIV
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other); Kilimanjaro Clinical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: EFV Kids
Record Dates: First submitted 2017-07-18; First posted 2017-07-24 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Efavirenz; Child Behavior; Cognitive Symptom; Medication Adherence; Drug-Related Side Effects and Adverse Reactions
Keywords: Efavirenz; Child Behavior; Cognition; Medication Adherence; Drug-Related Side Effects
MeSH Terms: conditions — Child Behavior; Neurobehavioral Manifestations; Medication Adherence; Drug-Related Side Effects and Adverse Reactions | interventions — efavirenz; Nevirapine; lopinavir-ritonavir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Efavirenz: Children using efavirenz-based cART for at least 6 months
  Interventions: Drug: Efavirenz
- Non-efavirenz: Children using non-efavirenz-based cART (nevirapine or Lopinavir-Ritonavir Drug Combination) for at least 6 months.
  Interventions: Drug: Nevirapine; Drug: Lopinavir-Ritonavir Drug Combination

INTERVENTIONS:
Drug: Efavirenz — Weight-based dosing according to the National Guidelines for the Management of HIV and AIDS
  Other Names: Efavirenz-group
  Groups: Efavirenz
Drug: Nevirapine — Weight-based dosing according to the National Guidelines for the Management of HIV and AIDS
  Other Names: Non-efavirenz group
  Groups: Non-efavirenz
Drug: Lopinavir-Ritonavir Drug Combination — Weight-based dosing according to the National Guidelines for the Management of HIV and AIDS
  Other Names: Non-efavirenz group
  Groups: Non-efavirenz

SUMMARY:
Efavirenz is among the preferred antiretroviral drugs for HIV-infected children. Increasing evidence shows that central nervous system side-effects in adults are more common than previously thought. Still, reliable data in children are lacking. As HIV-infected children nowadays have a prospect of reaching adulthood, there is an urgent need to identify potential long-term central nervous system side-effects, interfering with neurodevelopment and psychosocial maturation. Using validated tools, we assessed (1) competence (social/activities/school) and psychopathology (internalizing/externalizing problems), (2) cognitive performance (intelligence and working memory), and (3) adherence in Tanzanian children on an efavirenz or non-efavirenz based regimen

In this cross-sectional observational study the investigators will examine neuropsychiatric and neurocognitive functioning in 126 children (aged 6-11 years) on long-term combination antiretroviral therapy (cART) with or without efavirenz.

DETAILED DESCRIPTION:
In this cross-sectional observational study, we include HIV-infected children (6-12 years) on cART for ≥ 6 months, with viral loads ≤ 1000 copies/ml in Kilimanjaro Region, Tanzania. Psychopathology and competence will be assessed using the Child Behaviour Checklist. Cognitive performance will be assessed using the Raven's Coloured Progressive Matrices and the digit span test. Non-adherence is defined as any reported missed doses over the previous 3 days or <100% adherence since the last clinical visit. Analysis of covariance and logistic regression models will be used to assess differences between groups. .

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 until 12 years
* HIV seropositive
* Using cART, with or without efavirenz, for at least 6 months
* Registered patient at one of the participating centres
* In the presence of at least one parent or caregiver who is part if the child's life/upbringing

Exclusion Criteria:

* Switch of cART regimen in the last 6 months
* History of brain injury, mental health and cognitive impairment before starting cART
* HIV RNA >1000 copies/mL within the past year
* Any AIDS-defining illness or acute illness (e.g. fever, lowered consciousness, dehydration) at time of inclusion
* Children with parent(s) or caregiver(s) not wanting or not able to give informed consent

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Tanzanian children (6-12 years) living with HIV and receiving cART
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Neuropsychological symptoms: competence and psychopathology (internalizing/externalizing symptoms) | At day of inclusion
  Neuropsychological symptoms will be assessed using the Swahili version of the Child Behavior Checklist for 6-18 years (CBCL6-18)

SECONDARY OUTCOMES:
Cognitive functioning - non-verbal cognitive ability (general intelligence) | At day of inclusion
  Non-verbal cognitive ability will be assessed using the Raven's Progressive Matrices
Cognitive functioning - working memory | At day of inclusion
  Working memory will be assessed using the Wechsler Intelligence Scale for Children (WISC-III) Digit Span Test
Treatment adherence | At day of inclusion
  Treatment adherence will be measured using an adherence questionnaire, adapted from the PENTA 16 trial (permission obtained from the author prof. Giaquinto)

OTHER OUTCOMES:
Central nervous system symptoms | At day of inclusion
  The presence of central nervous system symptoms (yes/no) in the week prior to study visit will be assessed using a checklist composed of symptoms that have been linked to efavirenz in literature.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Kinabo, MD, PhD, Principal Investigator — Kilimanjaro Christian Medical Centre; André van der Ven, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (6):
- Tanzania (6):
  - Kilimanjaro Christian Medical Centre, Moshi, Kilimanjaro
  - Mawenzi Regional Hospital, Moshi, Kilimanjaro
  - Kibosho Hospital, Kibosho
  - Kiboroloni Dispensary, Moshi
  - Majengo Health Centre, Moshi
  - Pasua Health Centre, Moshi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van de Wijer L, Schellekens AFA, Burger DM, Homberg JR, de Mast Q, van der Ven AJAM. Rethinking the risk-benefit ratio of efavirenz in HIV-infected children. Lancet Infect Dis. 2016 May;16(5):e76-e81. doi: 10.1016/S1473-3099(16)00117-1. Epub 2016 Apr 18. PMID 27599655
- [Background] Mothapo KM, Schellekens A, van Crevel R, Keuter M, Grintjes-Huisman K, Koopmans P, van der Ven A. Improvement of Depression and Anxiety After Discontinuation of Long- Term Efavirenz Treatment. CNS Neurol Disord Drug Targets. 2015;14(6):811-8. doi: 10.2174/1871527314666150325235847. PMID 25808896
- [Background] Van de Wijer L, Kinabo GD, Mchaile DN, de Mast Q, Schellekens AFA, van der Ven AJAM. Safety Evaluation of Efavirenz in Children: Don't Forget the Central Nervous System. Clin Infect Dis. 2018 Mar 19;66(7):1150. doi: 10.1093/cid/cix926. No abstract available. PMID 29088326
- [Derived] Van de Wijer L, Mchaile DN, de Mast Q, Mmbaga BT, Rommelse NNJ, Duinmaijer A, van der Ven AJAM, Schellekens AFA, Kinabo GD. Neuropsychiatric symptoms in Tanzanian HIV-infected children receiving long-term efavirenz treatment: a multicentre, cross-sectional, observational study. Lancet HIV. 2019 Apr;6(4):e250-e258. doi: 10.1016/S2352-3018(18)30329-1. Epub 2019 Feb 12. PMID 30770324